CLINICAL TRIAL: NCT07094269
Title: Protocol for a Superiority Randomized Controlled Trial of a Group-Based Fatigue Management Program Versus Standard Information to Improve Self-Efficacy in Energy Conservation in Parkinson's Disease
Brief Title: Protocol of the Packer Managing Fatigue Program Versus Standard Information to Improve Energy Conservation Self-Efficacy in Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universita degli Studi di Genova (Other)
Responsible Party: Principal Investigator, Elisa Pelosin, Prof., Universita degli Studi di Genova
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: USGenova
Record Dates: First submitted 2025-07-22; First posted 2025-07-30 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: PARKINSON DISEASE (Disorder)
Keywords: occupational therapy; fatigue; parkinson's disease; self-management
MeSH Terms: conditions — Parkinson Disease; Fatigue

STUDY DESIGN:
Intervention Model Description: This will be a two-arm controlled trial adopting a superiority framework. Participants will be allocated to either the intervention group or the control group using a stratified block allocation approach with a 1:1 ratio.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Due to the nature of the intervention, neither participants nor care providers will be masked to treatment allocation. However, data analysts and outcome assessors responsible for evaluating clinician-reported outcomes will be masked to group assignment to reduce the risk of assessment bias. To ensure assessor blinding, the individuals performing clinical outcome evaluations were not involved in participant enrollment or intervention delivery and were not informed of the assigned treatment groups. Participants and staff were instructed not to disclose allocation information during assessments. No blinding procedures were applied to the appearance or labeling of interventions, as blinding was not feasible for other roles
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Packer Managing Fatigue Program (Experimental): Packer Managing Fatigue Group Program, delivered in groups of 8-10 by a licensed occupational therapist. The intervention will consist of six weekly sessions, each lasting 120 minutes, held in a dedicated outpatient room equipped with a whiteboard, group seating, and educational materials.
  Each session will address a specific theme: (1) The importance of Rest, (2) Communication and Body Mechanics, (3) Tools, Technology, and ergonomics, (4) Priorities and Standard (5) Putting it all Together, (6) Some Closing Thoughts. Materials will include a participant workbook2, printed handouts, pens, markers, and name tags. All materials will be provided in Italian. A structured intervention manual and session-specific checklists will guide therapist and ensure intervention fidelity.
  Interventions: Other: Occupational Therapy Intervention
- Fact sheets about Parkinson's disease (Placebo Comparator): Participants in the control group will be provided with six fact sheets (one per week) addressing general information about Parkinson's disease,. The control group reflects current standard care, as no structured fatigue intervention is routinely provided in this clinical setting.
  Interventions: Behavioral: Fact-sheets

INTERVENTIONS:
Other: Occupational Therapy Intervention — Participants in the intervention group will take part in the structured, manualized Packer Managing Fatigue Group Program (Packer et al.), delivered in groups of 8-10 by a licensed occupational therapist. The intervention will consist of six weekly sessions, each lasting 120 minutes, held in a dedicated outpatient room equipped with a whiteboard, group seating, and educational materials.
  Each session will address a specific theme: (1) The importance of Rest, (2) Communication and Body Mechanics, (3) Tools, Technology, and ergonomics, (4) Priorities and Standard (5) Putting it all Together, (6) Some Closing Thoughts. Materials will include a participant workbook2, printed handouts, pens, markers, and name tags. All materials will be provided in Italian.
  Arms: Packer Managing Fatigue Program
Behavioral: Fact-sheets — Participants in the control group will receive six weekly fact sheets containing general information about Parkinson's disease. These fact sheets serve as a placebo intervention to control for attention and information exposure, without providing any structured fatigue management strategies. This approach helps isolate the specific effects of the active intervention compared to usual care.
  Arms: Fact sheets about Parkinson's disease

SUMMARY:
This protocol describes a randomized, controlled, parallel-group, trial evaluating the effectiveness of a group-based fatigue management program for people with Parkinson's disease. The study will be conducted in Italy, with participant recruitment planned to begin on July 1st, 2025. The primary sponsor is the Department of Neuroscience, Rehabilitation, Ophthalmology, Genetics and Maternal Child Health (DINOGMI) at the University of Genoa, Italy. No external sources of monetary or material support have been declared. The study has received ethical approval from the University of Genoa's Research Ethics Committee (Comitato Etico per la Ricerca di Ateneo - CERA), under protocol number 2025.36, approved on April 3rd, 2025.

The scientific title of the trial is: Protocol for a Superiority Randomized Controlled Trial of a Group-Based Fatigue Management Program Versus Standard Information to Improve Self-Efficacy in Energy Conservation in Parkinson's Disease". The public title is: "Energy Matters: A Protocol of a Randomized Controlled Trial of a Group-Based Fatigue Management Program for People with Parkinson's Disease".

The study targets individuals diagnosed with idiopathic Parkinson's disease, experiencing fatigue. Eligible participants must be over 18 years old, present with Hoehn and Yahr stage ≤3.5, and score ≥4 on the Fatigue Severity Scale (FSS). Exclusion criteria include a Montreal Cognitive Assessment (MOCA) score below 21, presence of severe psychiatric comorbidities, medical conditions contributing independently to fatigue, inability to participate in group sessions, or involvement in other structured fatigue management programs.

Participants will be randomly allocated to one of two arms. The intervention group will attend a six-week Packer Managing Fatigue Program1 Sessions will be conducted in groups of 8-10 participants, led by a licensed occupational therapist. Topics covered include rest, communication, body mechanics, ergonomics, energy-conserving tools, prioritization, lifestyle balance, and goal setting. Sessions will use standardized materials such as participant workbooks2 and visual aids and will take place in appropriately equipped rooms. If a participant is absent from a scheduled group session for personal reasons, the occupational therapist will organize an individual make-up session before the next scheduled group session. This individual session will follow the same content and structure as the missed group session, based on the Packer Managing Fatigue Program. Its purpose is to ensure continuity and fidelity to the intervention, and to allow participants to stay aligned with the group program.

Participants in the control group will be provided with six fact sheets addressing general information about Parkinson's disease.

The primary outcome is the change in self-efficacy for performing energy conservation strategies, measured using the Self-Efficacy for Performing Energy Conservation Strategies Assessment (SEPECSA), assessed at baseline, post-intervention, and at a 3-month follow-up.

Secondary outcomes include measures of motor and non-motor symptoms (Movement Disorder Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Parts I and II), fatigue severity (Fatigue Severity Scale, Parkinson Fatigue Scale), Fatigue Impact (Modified Fatigue Impact Scale), quality of life (Parkinson Disease Questionnaire-39), participation and autonomy (Impact on Participation and Autonomy questionnaire), psychiatric symptoms (Hospital Anxiety and Depression Scale), and sleep disturbance (Pittsburgh Sleep Quality Index - PSQI). All outcomes will be reassessed immediately and 3 months after the end of the intervention.

The total planned sample size is 74 participants, with 37 individuals in each study arm.

For public queries, the contact person is Dr. Elisa Pelosin, Associate Professor at DINOGMI, University of Genoa (email: elisa.pelosin@unige.it). For scientific queries, the reference contact is the University of Genoa's Ethics Committee (email: presidente.cera@unige.it).

An individual participant data sharing plan is in place. As part of the informed consent process, participants will be asked whether they agree to allow their anonymized data to be shared for future research purposes. Only data from participants who provide explicit consent will be shared. Anonymized individual data will be made available upon reasonable request, in accordance with institutional policies and data protection regulations. Access will be granted by the corresponding author after publication and will remain open for five years

DETAILED DESCRIPTION:
Introduction

Fatigue is one of the most prevalent and disabling non-motor symptoms in Parkinson's disease (PD), affecting approximately 50% of individuals and significantly impairing occupational performance, participation in daily life, and overall quality of life. According to the systematic review and meta-analysis by Siciliano et al. (2018), fatigue in PD represents a frequent and distinct clinical feature that is not attributable to pharmacological side effects or comorbid psychiatric disorders. It can emerge in the early stages of the disease and tends to persist or worsen over time. As described by Friedman (2015), PD-related fatigue is characterized by a subjective sense of exhaustion and reduced energy, disproportionate to effort, unrelieved by rest, and affecting both physical and cognitive functioning. Its multidimensional and persistent nature makes it particularly difficult to treat.

Despite its considerable impact, no pharmacological treatments have demonstrated consistent efficacy for fatigue in PD. As a result, growing attention has been directed toward non-pharmacological approaches, particularly those delivered by occupational therapists. Occupational therapy interventions often focus on fatigue self-management and energy conservation strategies, aiming to support individuals in maintaining engagement in meaningful activities and improving daily functioning.

In this context, the Packer Managing Fatigue Group Program (MFGP) represents a structured, evidence-based occupational therapy intervention that has demonstrated effectiveness in populations with multiple sclerosis and post-polio syndrome. As highlighted in the systematic review by Kim et al. (2021), seven out of ten energy conservation studies were based on the MFGP, confirming it as one of the most evidence-supported interventions in the field. No adverse effects have been reported in previous studies evaluating the MFGP in other neurological populations.

Nonetheless, evidence supporting the use of the MFGPMFGP in individuals with PD remains extremely limited. To date, only one randomized controlled trial has been planned in this population. The protocol published by Alizadeh et al. (2022) describes the implementation of an individual, telehealth-based version of the program. While this study confirms the feasibility of a one-to-one delivery model, it does not examine the original group-based format, which has been shown to be cost-effective, socially engaging, and scalable in other clinical populations. Furthermore, participants in that study were drawn from heterogeneous diagnostic groups, and outcomes specific to individuals with PD were not reported separately.

Implementing the program in a group setting may enhance its therapeutic value by promoting peer support, shared learning experiences, and a sense of mutual accountability-factors that are known to facilitate sustained engagement in self-management behaviors.

Given the current lack of established treatment protocols for fatigue in Parkinson's disease, and the absence of evidence supporting even the individual delivery of the MFGP in this population, a comparator reflecting usual care was deemed most appropriate. At present, individuals with PD do not routinely receive targeted interventions for fatigue within standard clinical practice. Therefore, the control group in this study will receive a set of educational brochures specifically developed to provide structured, evidence-informed information about fatigue and energy conservation strategies. This approach ensures that all participants have access to relevant health information while allowing the study to assess the added value of structured, therapist-led group intervention over passive information provision.

Given the high prevalence of fatigue in PD, the lack of effective treatments, and the limited availability of standardized occupational therapy programs addressing this issue in Italy, there is a compelling need for further investigation. The objective of this trial is to evaluate the efficacy of the Packer Managing Fatigue Group Program, , in improving self-efficacy for energy conservation strategies in individuals with Parkinson's disease. Participants in the control group will be provided with six fact sheets addressing general information about Parkinson's disease. The primary outcome is self-efficacy, measured using the Self-Efficacy for Performing Energy Conservation Strategies Assessment (SEPECSA), with assessments conducted at baseline, immediately post-intervention, and at 3-month follow-up. This randomized controlled trial aims to determine whether the structured group program leads to superior outcomes compared to passive information delivery. This study addresses an unmet rehabilitative need and has the potential to inform future clinical guidelines for managing fatigue in PD through occupational therapy.

Methods

Patient and public involvement

Patients or members of the public were not involved in the initial design or development of this trial. The research questions, outcome measures, and intervention content were established based on clinical expertise, existing research evidence, and international best practices in occupational therapy for fatigue management. Nevertheless, the study team recognizes the value of incorporating patient perspectives and plans to engage participants during later stages of the research. Specifically, participants will be invited to: provide qualitative feedback on the acceptability and clarity of the intervention materials following the program, and contribute to the creation of a plain language summary of the trial results, ensuring it is accessible and meaningful for people living with Parkinson's disease.

Trial Design

This will be a two-arm controlled trial adopting a superiority framework. Participants were will be allocated to either the intervention group or the control group using a stratified block allocation approach with a 1:1 ratio.

Trial Setting

The trial will be conducted at a single site in Genoa, Italy, within the outpatient setting of the Neurology Clinic at the Department of Clinical and Experimental Neurosciences (DINOGMI), University of Genoa. The clinic is located near the main university hospital and functions as a tertiary care ambulatory center for individuals with neurological disorders. All participant recruitment, intervention delivery, and follow-up assessments will be conducted within this outpatient facility.

Eligibility Criteria

Participants were will be eligible for inclusion if they were are adults (aged >18 years) with a diagnosis of idiopathic PD, Hoehn and Yahr stage ≤3.5, a score ≥4 on the Fatigue Severity Scale (FSS), and a Montreal Cognitive Assessment (MoCA) score >221. Exclusion criteria included the presence of significant cognitive impairment, comorbid medical conditions that could independently contribute to fatigue, parkinsonism, non parlare fluentemente la lingua italianaor not being fluent in the Italian language, or an inability to participate in group-based sessions. Recruitment will be conducted through both neurologist referral and self-selection. In the referral pathway, clinicians will recommended participation during routine outpatient consultations at the Neurology Clinic Recruitment will occur through both neurologist referral and self-selection. In the referral pathway, neurologists will provide eligible patients with written information about the study during routine outpatient visits. Patients who express interest will be invited to contact the research team independently. Additionally, informational brochures will be distributed in Parkinson's associations and community clinics to support self-referral. For self-selection, informational brochures describing the study were will be distributed in Parkinson's clinics and centres across the region, including through the Ligure Parkinson Association For self-selection, informational brochures describing the study werewill be distributed at the Department of Neuroscience, Rehabilitation, Ophthalmology, Genetics and Maternal Child Health. Copies of recruitment materials are provided in the Supplementary Materials. As the trial will be conducted at a single site, no specific eligibility criteria for site selection were applied beyond the availability of suitable facilities for group-based interventions and follow-up assessments.

The intervention will be delivered by a licensed occupational therapist with clinical experience in neurological rehabilitation and be trained and licensed to deliver formal training in the Packer Managing Fatigue Group Program (MFGP) protocol. Prior to the trial, the therapist will completeed a standardized training and a familiarization process to ensure fidelity to the original intervention model.

Methods

Patient and public involvement, trial design

Patients wereill be actively involved at all stages of the trial, including its design, conduct, and dissemination, in accordance with established recommendations. During the initial design phase, approximately twenty individuals with Parkinson's disease were consulted to assess the perceived usefulness of a similar self-management fatigue group and to explore their expectations regarding meaningful improvements; this qualitative inquiry informed the identification of relevant outcomes. Throughout the intervention in the qualitative study, verbal feedback wasill be solicited from participants during each session and at the post-treatment assessment; all responses wereill be audio-recorded and fully transcribed by the researcher . Upon completion of the trial, a lay summary written in accessible language will be prepared and disseminated to all participants to communicate the study findings.

No changes were made to the trial protocol after commencement. The randomisation approach, eligibility criteria, intervention procedures, outcome measures (including methods of assessment and timepoints), target sample size, number of trial arms, duration of follow-up, and statistical analysis plan remained consistent with the pre-specified protocol. No unplanned or post hoc outcomes were introduced, and no modifications to trial conduct (e.g., site exclusion or adjustment of procedures) were required throughout the study period.

Participants, interventions, and outcomes

Participants in the intervention group will take part in thea structured, manualized fatigue self-management program based on the Packer Managing Fatigue Group Program, delivered in groups of 8-10 by a licensed occupational therapist. The intervention will consist of six weekly sessions, each lasting 120 minutes , held in a dedicated outpatient room equipped with a whiteboard, group seating, and educational materials.

Each session will address a specific theme: (1) rest and sleepThe importance of Rest, (2) Ccommunication and Bbody Mmechanics, (3) energy-conserving tTools, Technology, and ergonomics, (4) Priorities and Standard (5) Putting it all Together, prioritization, (5) lifestyle balance, and (6) goal settin(6) Some Closing Thoughts. Materials will include a participantparticipant workbook, printed handouts, pens, markers, and name tags. All materials will be provided in Italian. A structured intervention manual and session-specific checklists will guide therapists and ensure intervention fidelity.

The program will follow a standardized format without individual tailoring, although participants will be allowed to contact the therapist between sessions for clarification. Missed sessions will be rescheduled individually when feasible. The program will follow a standardized format in terms of structure and content; however, participants will be encouraged to personalize their between-session activities and homework based on their individual goals and routines. While session content will not be tailored, participants may contact the therapist between sessions for clarification. If a session is missed, an individual make-up session will be scheduled when feasible to ensure continuity.

The comparator group will receive six weekly brochures summarizing the same thematic content as the intervention group. These brochures will be delivered without interaction or facilitation. Both groups will receive identical written materials to ensure equivalence in informational exposure. The control group reflects current standard care, as no structured fatigue intervention is routinely provided in this clinical setting. Participants in the control group will receive six weekly fact sheets containing general information about Parkinson's disease. These fact sheets serve as a placebo intervention to control for attention and information exposure, without providing any structured fatigue management strategies. This approach helps isolate the specific effects of the active intervention compared to usual care. Participation in other psychoeducational or self-efficacy-based programs will be prohibited during the study period. Starting new physiotherapy or exercise programs will also not be allowed, although existing regimens may continue. Any new treatments or changes to ongoing regimens, including medications, physiotherapy, or structured exercise, will be systematically tracked and documented at each assessment point. This information will be considered in data analysis to control for potential confounding effects.

Participants may withdraw from the study at any time without justification or reprecussioin. If a participant is unable to continue attending sessions due to clinical worsening, caregiver burden, or logistical issues, the intervention will be discontinued, and no further sessions will be scheduled. In the event of adverse effects, distress, or significant decline in health status, discontinuation will be considered after clinical evaluation. No modifications to the intervention content or format will be implemented during the trial.

Adherence attendance will be monitored through attendance logs. Participants attending at least five of six sessions will be considered "treated as planned." To enhance adherence, reminder messages (SMS or phone call) will be sent the day before each session. Therapist adherence to the intervention will be ensured through comprehensive training prior to trial initiation, the use of a structured intervention manuals, and session-specific checklists developed by the principal investigator based on the manual. Therapists will be required to consult these checklists during the delivery of the intervention to ensure complete and accurate implementation of the prescribed procedures. Implementation fidelity will be ensured through comprehensive therapist training prior to trial initiation, the use of a structured intervention manual, and session-specific checklists developed based on the Managing Fatigue Program. At the end of each group session, therapist will complete the checklist to confirm which components were delivered. These data will be used to calculate a fidelity score (percentage of components delivered per session).

While receipt fidelity will not be formally tested, it will be supported through discussion, group reflection, and participant questions during sessions.

Enactment fidelity will be explored indirectly through follow-up assessments and participant-reported implementation of fatigue management techniques.

Participation in other fatigue-related or psychoeducational interventions will not be allowed during the study. The initiation of new physiotherapy or physical activity programs will also be restricted, as existing literature demonstrates the efficacy of physical activity in modulating the perception of fatigue impact, which could confound the study outcomes. Ongoing treatments may continue and will be documented at baseline and monitored throughout the trial. Any significant changes in concomitant care will be systematically recorded.

The primary outcome of the trial will be self-efficacy in applying energy conservation strategies, assessed using the SEPECSA. This instrument measures individuals' confidence in implementing specific fatigue management techniques in daily life.

Secondary outcomes will include: Perceived fatigue severity and impact, measured through the Fatigue Severity Scale (FSS), the Modified Fatigue Impact Scale (MFIS), and the Parkinson Fatigue Scale (PFS); Quality of life, assessed by the Parkinson's Disease Questionnaire-39 (PDQ-39); Participation and autonomy, measured using the Impact on Participation and Autonomy (IPA) and the Community Integration Questionnaire-Revised (CIQ-R); Sleep quality, assessed with the Pittsburgh Sleep Quality Index (PSQI); Emotional symptoms, evaluated using the Hospital Anxiety and Depression Scale (HADS) and Motor and non-motor symptoms, assessed through the Movement Disorder Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part I and II.

All outcomes will be assessed at three time points: baseline (T0), immediately post-intervention (T1), and three-month follow-up (T2).

All measures will be collected through self-reported questionnaires completed by participants using standardized and validated instruments. The outcomes have been selected based on clinical relevance and prior use in trials involving fatigue and Parkinson's disease. No formal core outcome set will be applied.

Given the non-invasive and behavioral nature of the intervention, no specific harms will be anticipated. Harms will be assessed through non-systematic, passive surveillance. At each group session and during the post-intervention (T1) and 3-month follow-up (T2) assessments, participants will be invited to spontaneously report any adverse events, discomfort, or difficulties related to the program.

These reports will be collected verbally by the occupational therapist referring neurologist delivering the intervention, who will not be blinded to group allocation. No formal coding system or severity grading scale will be used. Instead, any reported harmsharm will be recorded descriptively, including the nature of the event, its timing, and the participant's perception of its relationship to the intervention. These reports will be discussed with the principal investigator for clinical judgment and documentation.

The study will follow a three-phase timeline: (1) enrollment and screening, (2) intervention period, and (3) follow-up. The overall duration for each participant will be approximately 19 weeks, including baseline assessment, the 6-week intervention period, and a 3-month follow-up. After eligibility screening and informed consent (T-1 to T0), participants will undergo baseline assessments and be randomized into the intervention or comparator group (T0). The intervention or control materials will then be delivered weekly for six consecutive weeks (T1-T6). Outcome assessments will be conducted immediately after the intervention (T7) and again at 3-month follow-up (T19).

The sample size calculation for this trial was based on the primary outcome, namely the SEPECSA. As no previous study has used the SEPECSA in people with PD, the investigator consulted existing occupational therapy literature where the SEPECSA was used in populations with similar fatigue-related challenges. Based on these sources, the investigator assumed a moderate effect size (Cohen's d = 0.5) between the intervention and control groups.

Using this assumption and setting the type I error (α) at 0.05 and the type II error (β) at 0.20 (corresponding to 80% statistical power), the investigator performed a sample size calculation for a two-tailed independent samples t-test. The calculation indicated that a minimum of 65 participants (32.5 per group) would be required to detect a between-group difference of medium effect size at post-intervention. To account for potential attrition or loss to follow-up, estimated conservatively at 15% based on similar behavioral intervention studies in PD, the sample size was increased. The final target sample size will be 74 participants, with 37 participants per arm. The sample size calculation was performed using G*Power software version 3.1.9.7.

To ensure adequate participant enrollment and achieve the planned sample target, several recruitment strategies have been planned. Informational brochures distributed in healthcare facilities and specialized centers will be used, along with social media campaigns to increase the visibility of the study and reach a wider audience.

Assignment of interventions

The randomisation sequence will be computer-generated by an independent statistician using a computerized random number generator with randomly permuted blocks of equal length, each containing a fixed number of treatment allocations to balance enrolments over time using . The blocks will be stratified by cognitive status (MoCA scores between 21-26 and 27-30) to ensure balance across study groups. The randomisation sequence will be computer-generated by an independent statistician using a computerized random number generator with randomly permuted blocks of equal length. As soon as each block of 20 participants is recruited, they will be allocated to treatment groups to balance enrolments over time. The blocks will be stratified by cognitive status (MoCA scores between 22-26 and 28-31) to ensure balance across study groups within each block.

The allocation sequence will be concealed using sequentially numbered, opaque, sealed envelopes to prevent selection bias.

Separate intervention and assessment teams will be used. All assessment staff will be blinded to participant randomisation assignments. The personnel responsible for enrolling participants and assigning interventions will have no access to the random allocation sequence, which will be securely stored by A.B..

The randomisation sequence was computer generated using randomly permuted blocks of equal length each with fixed numbers of treatment allotments to balance enrolments over time. The blocks were stratified by Cognitive status (MOCA between 21-26 and 26-30) to ensure balance across the study groups. There were separate intervention and assessment teams and all assessment staff were blinded to participant randomisation assignment.

This study is an open-label trial. Due to the nature of the intervention, neither participants nor care providers nor data analysts were will be masked blinded to treatment allocation. However, data analysts and outcome assessors responsible for evaluating clinician-reported outcomes were will be masked blinded to group assignment in order toto reduce the risk of assessment bias. To ensure assessor blinding, the individuals performing clinical outcome evaluations were not involved in participant enrollment or intervention delivery and were not informed of the assigned treatment groups. Participants and staff were instructed not to disclose allocation information during assessments. No blinding procedures were applied to the appearance or labeling of interventions, as blinding was not feasible for other roles Data collection, management, and analysis Primary and secondary outcomes will be assessed by trained evaluators using clinician-reported outcome measures (MDS-UPDRS and MoCA) and self-report questionnaires, depending on the variable. Where applicable, instruments with established reliability and validity in the target population will be used.

Data will be collected on paper-based forms and subsequently entered into a secure electronic database. To ensure data quality, assessors will undergowent standardized training. Range checks, skip patterns, and internal consistency checks were will be built into the database to detect potential entry errors. Data collection forms are available upon request.

For participants who deviate from the protocol or withdraw, available outcome data will still be collected whenever possible. Reasons for non-adherence or withdrawal will be recorded systematically.

If the data are normally distributed, primary and secondary outcome comparisons between intervention and control groups will be conducted using repeated measures Repeated-Measure ANOVA (RM-ANOVA); otherwise, non-parametric alternatives will be used. Results will be reported with corresponding 95% confidence intervals and a significance level of p = 0.05. Primary and secondary outcomes will be analyzed using linear mixed-effects models (LMMs) to assess differences between intervention and control groups over the three time points (T0, T1, T2). Baseline values (T0) will be included as covariates to control for initial differences. Random effects will account for within-subject correlations across time. If model assumptions are violated or data are not normally distributed, generalized linear mixed models (GLMMs) with appropriate link functions will be employed. Results will be reported with 95% confidence intervals and a significance level of p = 0.05.

All participants will be included in the intention-to-treat (ITT) analysis. Modified ITT analysis will include all randomized participants who completed at least five of six sessions Modified ITT analysis will include all randomized participants with at least one post-baseline assessment. Completion of treatment will be defined as attendance at five of six sessions. Per-protocol analysis will include participants who adhered to the treatment protocol. The safety set includes data collected from participants who received at least one intervention after randomization and for whom safety indicators were documented. Primary analyses will be conducted using multiple imputation methods for missing observations at baseline, post-intervention, and at follow-up, assuming missing data are missing at random.l. Missing data at the item level within questionnaires will be handled according to standard scoring procedures, including mean substitution when appropriate. For missing observations at baseline, post-intervention, and follow-up (i.e., entire missing assessments), multiple imputation methods will be used, assuming data are missing at random. Multiple imputation is preferred over mean substitution for missing assessments because it provides less biased estimates and better accounts for the uncertainty due to missing data. Prespecified sensitivity analyses will be conducted for all participants using complete-case data at each time point.

Subgroup analyses will explore the potential moderating effect of baseline characteristics such as age group (<65 vs ≥65), cognitive status or sex, using interaction terms in regression models. Sensitivity analyses will examine the impact of protocol deviations and missing data assumptions.

ELIGIBILITY:
Inclusion Criteria:

* aged >18 years
* diagnosis of idiopathic Parkinson's disease (PD)
* Hoehn and Yahr stage ≤3.5
* Fatigue Severity Scale (FSS) >= 4

Exclusion Criteria:

* Montreal Cognitive Assessment (MoCA) score <22
* comorbid medical conditions that could independently contribute to fatigue
* not being fluent in the Italian language
* Parkinsonism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Self-Efficacy for Performing Energy Conservation Strategies Assessment (SEPECSA) | Baseline, End of Treatment (7 week) and at 3 months
  The SEPECSA was originally developed by Liepold and Mathiowetz's (2005) confidence in applying energy conservation strategies among individuals with MS. It consists of 14 items listing energy-saving strategies, with each item scored on a 10-point Likert-type scale (1 = "I never do it," 10 = "I always do it"). The assessment took approximately 10-15 minutes to complete. The final score was found by adding the total items' score and dividing it by 14. Psychometric properties of the original SEPECSA include high internal consistency (Cronbach's alpha = 0.93) and acceptable construct validity, as demonstrated by its correlation with fatigue levels and quality-of-life measures. This instrument measures individuals' confidence in implementing specific fatigue management techniques in daily life.

SECONDARY OUTCOMES:
Fatigue Severity Scale (FSS) | Baseline, End of Treatment (7 week) and at 3 months
  Fatigue severity scale (FSS) is one of the most commonly used tools to measure fatigue. It was developed by Krupp et al. for patients with systemic lupus erythematosus and multiple sclerosis. However, it was later validated for various conditions such as obesity, chronic hepatitis C, cirrhosis, Parkinson's disease, postpartum, stroke, and post-polio. It was also validated into several languages such as Norwegian, Turkish, Swiss,German, English, Portuguese, Greek,Persian, Arabic, Italian, Chinese, Finnish,and Russian. The FSS is a 9-item self-reported scale. Each item is rated on a 7-point Likert scale from 1 = "strongly disagree" to 7 = "strongly agree". The total score is the unweighted mean of all items.
Parkinson Fatigue Scale (PFS) | Baselibe, End of Treatment /7 weeks) and 3 months
  The Parkinson Fatigue Scale (PFS) contains 16 questions: 7 questions related to tiredness and the effect of physical fatigue and 9 questions that evaluate the effect of fatigue on performance and daily activities. As mentioned, the questionnaire was completed by the subjects, and the score for each question ranged from 1 (definitely disagree) to 5 (definitely agree)
Modified Fatigue Impact Scale (MFIS) | Baseline, End of Treatment /7 weeks), 3 months
  The MFIS questionnaire is the modified form of the 40-item Fatigue Impact Scale (FIS) that has three dimensions and 21 questions (Fisk et al., 1994a). The total MFIS score is composed of nine items for physical status, 10 items for cognitive status, and two items for psychosocial function status.
Parkinson's Disease Questionnaire-39 (PDQ-39) | Baseline, End of Treatment (7 weeks), at 3 months
  The PDQ-39 comprises 39 questions with five different options of answer related to the frequency of the disease manifestation. Answers refer to impact of the illness on the PD patient's life in the previous month, as explained before the interview. The 39 questions are divided into 8 dimensions: mobility (1-10 questions), activities of daily living (ADL) (11-16 questions), emotional wellbeing (17-22 questions), stigma (23-26 questions), social support (27-29 questions), cognition (30-33 questions), communication (34-36 questions), and bodily discomfort(37-39 questions). The score for each question ranges from zero (0) to four (4): "never" = 0; "occasionally" = 1; "sometimes" = 2; "often" = 3; "always" = 4. The final score is the result of the following equation: the sum of each question score divided by the result times 4 (the maximal score for each question), divided by the total number of questions. This result is multiplied times by 100. Each dimension score ranges from 0 to 100.
Impact on Participation and Autonomy (IPA) | Baseline, end of treatment /7 weeks), at 3 months
  The IPA is a generic self-report outcome measure designed for use in adults with chronic health conditions. It examines several aspects of participation and autonomy through two different scales: IPA-I and IPA-II.
  IPA-I quantifies perceived limitations in participation and autonomy in relation to 32 different life situations across five subscales: autonomy indoors (7 items); family role (7 items); autonomy outdoors (5 items); social life and relationships (7 items); work and education (6 items). For each question there are 5 response options: 0-very good, 1-good, 2-fair, 3-poor, and 4-very poor.
  IPA-II examines the extent to which these limitations are experienced as problematic. This is evaluated with 9 items, which cover 9 different areas of participation and autonomy: mobility; self care; activities in and around the house; looking after money; leisure; social life and relationships; paid or voluntary work; education and training; helping and supporting other people. The perceive
Community Integration Questionnaire-Revised (CIQ-R) | Baseline, End of Treatment (7 weeks), at three months
  The CIQ-R is an 18-item questionnaire designed to be a brief, reliable measure of home, social, productivity integration, and electronic social networking, designed at first to be administered to people with TBI.
Pittsburgh Sleep Quality Index (PSQI) | Baseline, end of treatment /7 weeks), three months
  Pittsburgh Sleep Quality Index: The 19-item PSQI is the most used retrospective self-report questionnaire, which measures sleep quality over the previous month [18]. Seven clinically derived domains of sleep difficulties (sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction) are assessed by the questionnaire.
Hospital Anxiety and Depression Scale (HADS) | Baseline, end of treatment (7 weeks), at 3 months
  The HADS is a self-report rating scale of 14 items on a 4-point Likert scale (range 0-3). It is designed to measure anxiety and depression (7 items for each subscale). The total score is the sum of the 14 items, and for each subscale the score is the sum of the respective seven items (ranging from 0-21). It is worth noting that items referring to depression symptoms that describe somatic aspects of depression (e.g. insomnia and weight loss) are not included in the scale.
Movement Disorder Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part I and II | Baseline, end of Treatment (7 weeks), at 3 months
  Part I - Non-Motor Experiences of Daily Living focuses on symptoms not directly related to movement, such as sleep disturbances, mood changes, cognitive issues, and autonomic dysfunction. These are reported by the patient and reflect how non-motor symptoms affect everyday life.
  Part II - Motor Experiences of Daily Living addresses motor difficulties experienced in daily activities, including speech, walking, dressing, and eating. It captures the patient's perspective on how motor symptoms impact functional ability.
  Each item in both parts is rated on a scale from 0 to 4: 0 means normal; 1 (slight) indicates symptoms with no functional impact; 2 (mild) reflects modest impact; 3 (moderate) indicates considerable but not disabling effects; and 4 (severe) signifies that the symptom prevents function.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neuroscience, Rehabilitation, Ophthalmology, Genetics and Maternal Child Health (DINOGMI) University of Genoa Genoa, Italy, Genova, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Antonini A, Abbruzzese G, Ferini-Strambi L, Tilley B, Huang J, Stebbins GT, Goetz CG, Barone P; MDS-UPDRS Italian Validation Study Group; Bandettini di Poggio M, Fabbrini G, Di Stasio F, Tinazzi M, Bovi T, Ramat S, Meoni S, Pezzoli G, Canesi M, Martinelli P, Maria Scaglione CL, Rossi A, Tambasco N, Santangelo G, Picillo M, Morgante L, Morgante F, Quatrale R, Sensi M, Pilleri M, Biundo R, Nordera G, Caria A, Pacchetti C, Zangaglia R, Lopiano L, Zibetti M, Zappia M, Nicoletti A, Quattrone A, Salsone M, Cossu G, Murgia D, Albanese A, Del Sorbo F. Validation of the Italian version of the Movement Disorder Society--Unified Parkinson's Disease Rating Scale. Neurol Sci. 2013 May;34(5):683-7. doi: 10.1007/s10072-012-1112-z. Epub 2012 Jun 8. PMID 22678179
- [Background] Curcio G, Tempesta D, Scarlata S, Marzano C, Moroni F, Rossini PM, Ferrara M, De Gennaro L. Validity of the Italian version of the Pittsburgh Sleep Quality Index (PSQI). Neurol Sci. 2013 Apr;34(4):511-9. doi: 10.1007/s10072-012-1085-y. Epub 2012 Apr 13. PMID 22526760
- [Background] Franchignoni F, Ferriero G, Giordano A, Guglielmi V, Picco D. Rasch psychometric validation of the Impact on Participation and Autonomy questionnaire in people with Parkinson's disease. Eura Medicophys. 2007 Dec;43(4):451-61. PMID 18084167
- [Background] Pietrodarchi A, Berardi A, Galeoto G, Panuccio F, Simeon R. Validation of IPA and SEPECSA in Italian Individuals With Multiple Sclerosis: A Psychometric Study. OTJR (Thorofare N J). 2025 May 12:15394492251331445. doi: 10.1177/15394492251331445. Online ahead of print. PMID 40353487
- [Background] Galeoto G, Colalelli F, Massai P, Berardi A, Tofani M, Pierantozzi M, Servadio A, Fabbrini A, Fabbrini G. Quality of life in Parkinson's disease: Italian validation of the Parkinson's Disease Questionnaire (PDQ-39-IT). Neurol Sci. 2018 Nov;39(11):1903-1909. doi: 10.1007/s10072-018-3524-x. Epub 2018 Aug 7. PMID 30088166
- [Background] Finlayson M, Preissner K, Cho C. Outcome moderators of a fatigue management program for people with multiple sclerosis. Am J Occup Ther. 2012 Mar-Apr;66(2):187-97. doi: 10.5014/ajot.2012.003160. PMID 22394528
- [Background] Akbar N, Turpin K, Petrin J, Smyth P, Finlayson M. A pilot mixed-methods evaluation of MS INFoRm: a self-directed fatigue management resource for individuals with multiple sclerosis. Int J Rehabil Res. 2018 Jun;41(2):114-121. doi: 10.1097/MRR.0000000000000271. PMID 29324506
- [Background] Hersche R, Weise A, Michel G, Kesselring J, Bella SD, Barbero M, Kool J. Three-week inpatient energy management education (IEME) for persons with multiple sclerosis-related fatigue: Feasibility of a randomized clinical trial. Mult Scler Relat Disord. 2019 Oct;35:26-33. doi: 10.1016/j.msard.2019.06.034. Epub 2019 Jun 29. PMID 31280074
- [Background] Gamble C, Dudley L, Allam A, Bell P, Goodare H, Hanley B, Preston J, Walker A, Williamson P, Young B. Patient and public involvement in the early stages of clinical trial development: a systematic cohort investigation. BMJ Open. 2014 Jul 23;4(7):e005234. doi: 10.1136/bmjopen-2014-005234. PMID 25056972
- [Background] Thomas S, Thomas PW, Kersten P, Jones R, Green C, Nock A, Slingsby V, Smith AD, Baker R, Galvin KT, Hillier C. A pragmatic parallel arm multi-centre randomised controlled trial to assess the effectiveness and cost-effectiveness of a group-based fatigue management programme (FACETS) for people with multiple sclerosis. J Neurol Neurosurg Psychiatry. 2013 Oct;84(10):1092-9. doi: 10.1136/jnnp-2012-303816. Epub 2013 May 21. PMID 23695501
- [Background] Alizadeh N, Packer TL, Sturkenboom I, Eskes G, Warner G. Managing Fatigue in Parkinson's Disease: Protocol for a Pilot Randomized Controlled Trial. Can J Occup Ther. 2022 Jun;89(2):180-189. doi: 10.1177/00084174221085449. Epub 2022 Mar 15. PMID 35287487
- [Background] Packer, T.L., Lehman, M.J., Brink, N., & Sauriol, A. (2022). Packer Managing Fatigue: A Six-Week Self-Management Group Program (2nd ed., Participant Manual). Think Self-Management Inc. https://www.thinkselfmanagement.ca. ISBN: 978-1-7387441-0-7
- [Background] Packer, T.L., Lehman, M.J., Brink, N., & Sauriol, A. (2022). Packer Managing Fatigue: A Six-Week Self-Management Group Program (2nd ed., Therapist Manual). Think Self-Management Inc. https://www.thinkselfmanagement.ca. ISBN: 978-1-7387441-0-7